CLINICAL TRIAL: NCT01516086
Title: A 12-week Randomized, Multiple-Dose, Double-Blind, Placebo-Controlled, Parallel-Group Study to Replicate Efficacy of Nebulized Fluticasone Propionate (FP) in Adult Subjects With Partly Controlled and Uncontrolled Asthma
Brief Title: A 12-Week Study in Adult Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191-092
Record Dates: First submitted 2012-01-13; First posted 2012-01-24 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Asthma
Keywords: Controlled; uncontrolled
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Fluticasone Propionate (FP) - arm 1 (Experimental): FP BID (twice daily)
  Interventions: Drug: Fluticasone Propionate (FP)
- Fluticasone propionate (FP) - arm 2 (Experimental): FP BID
  Interventions: Drug: Fluticasone Propionate (FP)
- Fluticasone Propionate (FP) - arm 3 (Experimental): FP BID
  Interventions: Drug: Fluticasone Propionate (FP)
- FLuticasone Propionate (FP) - Arm 4 (Experimental): FP BID
  Interventions: Drug: Fluticasone Propionate (FP)
- Fluticasone Propionate (FP) - Arm 5 (Experimental): FP BID
  Interventions: Drug: Fluticasone Propionate (FP)
- Placebo - Arm 6 (Placebo Comparator): Placebo inhalation solution
  Interventions: Drug: Fluticasone Propionate (FP)

INTERVENTIONS:
Drug: Fluticasone Propionate (FP) — FP Inhalation BID
  Other Names: No other names applicable

SUMMARY:
This will be a multi-center, randomized, placebo controlled parallel-group study to Replicate Efficacy of Nebulized Fluticasone Propionate (FP) in Adult Subjects with Partly Controlled and Uncontrolled Asthma. Individual participation will be approximately 16 weeks, including 12 weeks of double-blind treatment.

DETAILED DESCRIPTION:
The primary outcome measure is FEV1 (Forced Expiry Volume in 1 second) and the secondary outcome measure is Peak Expiratory Flow Rate (PEFR), Asthma Control Questionnaire (ACQ), Nighttime awakenings and rescue medication usage.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated written informed consent form prior to the conduct of any study procedures
2. Males and females between ≥ 18 and ≤ 60 years old.
3. Non-smoker for at least 1 year prior to Visit 1, with a smoking history of no more than 10 pack-years (e.g., 1 pack [20 cigarettes] per day for 10 years).

6.Ability to understand and comply with the protocol requirements (including completion of daily PEFR, PFT and ACQ), instructions and protocol-stated restrictions.

7.Women of child-bearing potential (WOCBP) must have a negative pregnancy test at the screening visit. WOCBP include: any female who has experienced menarche and is not post-menopausal (defined as amenorrhea for at least 12 consecutive months), or has not undergone surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation). Women who are using acceptable contraceptive medications or devices to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy) will be considered WOCBP.

WOCBP must agree to avoid becoming pregnant for the duration of the study by using adequate contraception at study entry and throughout the trial. Examples of adequate contraception include the following:

* Norplant
* Medroxyprogesterone acetate injection
* Oral contraception
* Double-barrier method (e.g., condom and spermicide)
* Abstinence, with one of the above WOCBP will be advised to notify the Investigator of any changes in their pregnancy status or any change in contraceptive use.

  8.Agreement by subject to abide by the study protocol and its restrictions.

Exclusion Criteria:

1. Past or present disease, excluding asthma, which as judged by the investigator, may place the subject at increased risk of complications, interfere with study participation, or confound any of the study objectives These diseases include, but are not limited to cardiovascular disease, malignancy, gastrointestinal disease, hepatic disease, diabetes type I or uncontrolled diabetes, type II, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including, but not confined to chronic bronchitis, emphysema, bronchiectasis, COPD, eosinophilic bronchitis or pulmonary fibrosis).
2. An upper or lower respiratory tract infection within 4 weeks of Visit 1 and prior to Visit 2
3. A history of hypersensitivity to the study drug or its components, including albuterol as rescue medication.
4. History of illegal drug or alcohol abuse within the past 5 years.
5. Pregnant or lactating women.
6. Use of > 8 inhalations per day of SABA on any two consecutive days from screening to randomization (Visits 1 and 2).
7. Use of an investigational drug or device within 30 days prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 498 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
FEV1 (Forced Expiry Volume in 1 second) | FEV1 at Week 12

SECONDARY OUTCOMES:
Peak Expiratory Flow Rate (PEFR) | PEFR at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Imtiaz Chaudry, Study Director — Dey
Locations (1):
- CU Pharmaceutical Research, Rock Hill, South Carolina, United States